CLINICAL TRIAL: NCT00958789
Title: A Prospective, Post-market, Multi-center Study of the Outcomes of the Triathlon® Total Stabilizer (TS) Total Knee System
Brief Title: Triathlon Total Stabilizer (TS) Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triathlon TS Knee (Other): Triathlon TS Knee System
  Interventions: Device: Triathlon TS Knee System

INTERVENTIONS:
Device: Triathlon TS Knee System — Total knee replacement for revision cases

SUMMARY:
This study will be a prospective, non-randomized evaluation of the change between preoperative and postoperative outcomes for those receiving the Triathlon® TS Total Knee System for a revision knee operation. The mean total Knee Society Score (for pain, motion and function) change is not 10% worse than, or is superior to, the expected change according to published revision total knee replacement data, for cases implanted with the Triathlon® TS Total Knee System as compared from preoperative to 2 years postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an Institutional Review Board (IRB) approved, study specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female age 18 years or older at time of study device implantation.
* Patient is a candidate for revision of all femoral and tibial components of a total knee replacement.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) > 40.
* Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* Patient has a failed unicondylar knee prosthesis.
* Patient has a known sensitivity to device materials.
* Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-07; Primary Completion 2016-04-25 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirby D Hitt, M.D., Study Chair — Scott & White Hospital
Locations (12):
- United States (12):
  - The CORE Institute, Phoenix, Arizona
  - Heekin Institute for Orthopedic Research, Jacksonville, Florida
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Rothman Institute, Egg Harbor, New Jersey
  - Ridgewood Orthopedics, Ridgewood, New Jersey
  - Upstate Bone and Joint Center, East Syracuse, New York
  - University of North Carolina Orthopedics, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wellington Orthopaedic & Sports Medicine, Cincinnati, Ohio
  - The Orthopaedic Center, Tulsa, Oklahoma
  - Scott & White Clinic, Temple, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 226 participants/228 knees were enrolled in the study. 47 participants/47 knees were censored from the main cohort. One bilateral participant had one knee censored and one knee included in study so this participant counts in the total. Therefore, 180 participants/181 knees are followed and applicable data is reflected in this record.
Period: Overall Study
Arm/Group | Triathlon TS Knee
Started | 180
Completed (1 bilateral participant had a knee complete primary endpoint; other knee was revised) | 130 (Participant status at the 2 year primary outcome interval determined Completed/Not Completed counts.)
Not Completed | 50
Not completed — Death | 5
Not completed — Lost to Follow-up | 14
Not completed — Withdrawal by Subject | 17
Not completed — No 2 yr. Knee Society Score data | 4
Not completed — 2 yr. Knee Society Score not calculable | 1
Not completed — Subject terminated | 2
Not completed — Revision | 7

BASELINE CHARACTERISTICS:
Population: Participants who were censored are not included in baseline analysis.
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.25 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 81

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score (KSS) Change From Preoperative Time Point to 2 Years
Description: KSS Pain score, KSS Function score, Total Combined KSS
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
  Additionally, the KSS Pain subscore and KSS Function subscore are added together to obtain a total combined score (minimum score 0, maximum score 200).
Time Frame: pre-op, 2 years
Population: KSS Function Score at 2 years - One case had a calculable score for Function and not for Pain/Motion. Therefore, the case was not included in the Combined KSS Score and Participant Flow completed total of 130.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 177
Number analyzed (knees) | 178
units on a scale
  KSS Pain/motion score preoperative: number analyzed (Participants) | 169
  KSS Pain/motion score preoperative: number analyzed (knees) | 170
  KSS Pain/motion score preoperative | 39.81 (21.12)
  KSS Pain/motion score 2 yrs.: number analyzed (Participants) | 130
  KSS Pain/motion score 2 yrs.: number analyzed (knees) | 130
  KSS Pain/motion score 2 yrs. | 83.97 (15.95)
  KSS Function score preoperative | 41.43 (23.09)
  KSS Function score 2 yrs.: number analyzed (Participants) | 131
  KSS Function score 2 yrs.: number analyzed (knees) | 131
  KSS Function score 2 yrs. | 72.90 (25.12)
  Combined KSS score preoperative: number analyzed (Participants) | 169
  Combined KSS score preoperative: number analyzed (knees) | 170
  Combined KSS score preoperative | 82.96 (34.96)
  Combined KSS score 2 yrs.: number analyzed (Participants) | 130
  Combined KSS score 2 yrs.: number analyzed (knees) | 130
  Combined KSS score 2 yrs. | 157.05 (36.13)
Statistical Analysis 1: Comparison: Triathlon TS Knee; Test type: Non-Inferiority — For the primary efficacy hypothesis, H0, the total KSS change from preoperative to 2 years postoperative will be less than or equal to delta. The alternative hypothesis, Ha, will be that the total KSS change from preop to 2 years postoperative is greater than delta. When delta=63, the hypothesis will test for non-inferiority. When delta=70, the hypothesis will test for superiority. H0: mean 2-year - mean preop less than or equal to delta. Ha: mean 2-year - mean preop greater than delta; Mean Difference (Final Values) = 70.70, 95% CI 1-sided [lower limit 64.43]

2. Secondary Outcome: Knee Society Score (KSS) Functional Results Stratified by Joint Line Restoration Groups at 2 and 5 Years Postoperative
Description: This outcome measure shows the results of the KSS Functional Score for the groupings of the Joint Line Restoration (JLR). The 2 groups of JLR were stratified by the amount in mm that the joint line was restored to the physiological joint line postoperative. One group was those that were restored to ≤ 5 mm and the other was those that were restored to > 5mm.
  The Functional Score of the Knee Society Clinical Rating System ranges from a potential minimum score of 0 to a maximum score of 100 points. It is based on points assigned to ability to walk, climb stairs and the use of ambulatory aids. A higher value represents a better outcome.
Time Frame: 2 years, 5 years
Population: Data based on knees with available radiographic and clinical data at 2 years and 5 years postoperative.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Groups:
- Joint Line Restoration (JLR) ≤ 5 mm; Joint Line Restoration (JLR) > 5 mm: The Joint Line Restoration (JLR) is a measure in mm that the joint line was restored to the physiological joint line postoperative.
Arm/Group | Joint Line Restoration (JLR) ≤ 5 mm | Joint Line Restoration (JLR) > 5 mm
Number analyzed (Participants) | 49 | 32
Number analyzed (Knees) | 49 | 32
units on a scale
  KSS Function Score at 2yr | 75.31 (22.81) | 70.00 (25.02)
  KSS Function Score at 5yr: number analyzed (Participants) | 33 | 22
  KSS Function Score at 5yr: number analyzed (Knees) | 33 | 22
  KSS Function Score at 5yr | 66.82 (23.31) | 71.36 (26.78)

3. Secondary Outcome: Knee Stability Results Stratified by Joint Line Restoration Groups at 2 and 5 Year Postoperative
Description: Measures the knee stability results for the groupings of the Joint Line Restoration (JLR). The 2 groups of JLR were stratified by amount in mm that the joint line was restored to physiological joint line postoperative. One group were restored to ≤ 5 mm and the other were restored to > 5mm. Knee stability is evaluated in the anterior-posterior (AP) and medial-lateral (ML) planes.
  AP drawer test determines instability in mm of the tibia. It was done in the AP plane in both JLR groupings (≤ 5mm and > 5mm) at 2 years and 5 years. The AP measurements were sub categorized into 5mm and 5-10mm.
  ML is tested with a varus valgus stress test to determine any instability as measured in degrees. The ML measurements were done in both JLR groupings (≤ 5mm and > 5mm) at 2 years and 5 years with all results in only one category of < 5 degrees.
  The higher the number of degrees or mm measured the more instability in the knee.
Time Frame: 2 year and 5 year postoperative
Population: Data based on knees with available radiographic and clinical data at 2 years and 5 years postoperative.
Measure: Number; unit: Knees
Units Other Than Participants: Knees
Groups:
- Joint Line Restoration (JLR) > 5mm: The Joint Line Restoration (JLR) is a measure in mm that the joint line was restored to the physiological joint line postoperative.
Arm/Group | Joint Line Restoration (JLR) ≤ 5 mm | Joint Line Restoration (JLR) > 5mm
Number analyzed (Participants) | 49 | 32
Number analyzed (Knees) | 49 | 32
Knees
  Knee Stability AP < 5mm at 2 years | 47 | 29
  Knee Stability AP 5-10mm at 2 years | 2 | 3
  Knee Stability AP < 5mm at 5 years: number analyzed (Participants) | 31 | 22
  Knee Stability AP < 5mm at 5 years: number analyzed (Knees) | 31 | 22
  Knee Stability AP < 5mm at 5 years | 30 | 21
  Knee Stability AP 5-10mm at 5 years: number analyzed (Participants) | 31 | 22
  Knee Stability AP 5-10mm at 5 years: number analyzed (Knees) | 31 | 22
  Knee Stability AP 5-10mm at 5 years | 1 | 1
  Knee Stability ML< 5 degrees at 2 years | 49 | 32
  Knee Stability ML < 5 degrees at 5 years: number analyzed (Participants) | 31 | 22
  Knee Stability ML < 5 degrees at 5 years: number analyzed (Knees) | 31 | 22
  Knee Stability ML < 5 degrees at 5 years | 31 | 22

4. Secondary Outcome: Anterior Knee Pain Results Stratified by Joint Line Restoration Groups at 2 and 5 Years Postoperative
Description: Measures the presence or absence of anterior knee pain in the groupings of the Joint Line Restoration (JLR). The 2 groups of JLR were stratified by the amount in mm that the joint line was restored to the physiological joint line postoperative. One group was those that were restored to ≤ 5 mm and the other was those that were restored to > 5mm.
  Anterior knee pain is determined by clinical examination with patient and clinician whether it is present or absent.
Time Frame: 2 year and 5 year postoperative
Population: Data based on knees with available radiographic and clinical data at 2 years and 5 years postoperative. There was an one more anterior knee pain evaluation as compared to knee stability and KSS Function as there was one missing value on those two evaluations.
Measure: Number; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Joint Line Restoration (JLR) ≤ 5 mm | Joint Line Restoration (JLR) > 5 mm
Number analyzed (Participants) | 50 | 32
Number analyzed (Knees) | 50 | 32
Knees
  Anterior Knee Pain Absent at 2 yrs | 45 | 28
  Anterior Knee Pain Present at 2 yrs. | 5 | 4
  Anterior Knee Pain Absent at 5 yrs.: number analyzed (Participants) | 33 | 22
  Anterior Knee Pain Absent at 5 yrs.: number analyzed (Knees) | 33 | 22
  Anterior Knee Pain Absent at 5 yrs. | 26 | 20
  Anterior Knee Pain Present at 5 yrs.: number analyzed (Participants) | 33 | 22
  Anterior Knee Pain Present at 5 yrs.: number analyzed (Knees) | 33 | 22
  Anterior Knee Pain Present at 5 yrs. | 7 | 2

5. Secondary Outcome: Short Form Health Survey (SF-36) Health Survey Change From Pre-op to Post-op Visits
Description: The SF-36 Health Survey is a 36-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: pre-op, 1, 2, 5 years
Population: Participants/knees with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 178
Number analyzed (Knees) | 179
units on a scale
  SF-36 Physical Score Preoperative | 32.43 (8.07)
  SF-36 Physical Score 1 year: number analyzed (Participants) | 144
  SF-36 Physical Score 1 year: number analyzed (Knees) | 145
  SF-36 Physical Score 1 year | 41.30 (10.49)
  SF-36 Physical Score 2 year: number analyzed (Participants) | 133
  SF-36 Physical Score 2 year: number analyzed (Knees) | 133
  SF-36 Physical Score 2 year | 40.55 (11.60)
  SF-36 Physical Score 5 year: number analyzed (Participants) | 91
  SF-36 Physical Score 5 year: number analyzed (Knees) | 91
  SF-36 Physical Score 5 year | 38.42 (10.44)
  SF-36 Mental Score Preoperative | 45.85 (14.81)
  SF-36 Mental Score 1 year: number analyzed (Participants) | 144
  SF-36 Mental Score 1 year: number analyzed (Knees) | 145
  SF-36 Mental Score 1 year | 52.57 (12.33)
  SF-36 Mental Score 2 year: number analyzed (Participants) | 133
  SF-36 Mental Score 2 year: number analyzed (Knees) | 133
  SF-36 Mental Score 2 year | 52.42 (11.99)
  SF-36 Mental Score 5 years: number analyzed (Participants) | 91
  SF-36 Mental Score 5 years: number analyzed (Knees) | 91
  SF-36 Mental Score 5 years | 54.07 (11.81)

6. Secondary Outcome: Number of Knees With Radiographic Stability at 1, 2 and 5 Years Postoperative
Description: The scoring system was based on the Knee Society guidelines and determined by measuring the width of the radiolucent lines for each of the zones of the implant components in millimeters.
  The total widths are added for each zone which produces a numerical score. Radiolucency in at least 50% of a zone and measuring at least 1 mm in width is defined as radiolucency present. Failure is defined as a score of 10 or greater, regardless of symptoms and considered as radiographic instability.
Time Frame: 1, 2, 5 years
Population: Data based on knees with available data at 1, 2 and 5 years postoperative at the tibial and femoral component interface.
Measure: Number; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 148
Number analyzed (Knees) | 149
Knees
  Radiographically unstable at 1 year | 2
  Radiographically unstable at 2 year: number analyzed (Participants) | 129
  Radiographically unstable at 2 year: number analyzed (Knees) | 129
  Radiographically unstable at 2 year | 0
  Radiographically unstable at 5 year: number analyzed (Participants) | 80
  Radiographically unstable at 5 year: number analyzed (Knees) | 80
  Radiographically unstable at 5 year | 0

7. Secondary Outcome: Number of Knees With a Revision of Femoral and/or Tibial Baseplate Component
Description: Revision was defined as the removal of either the femoral component or the tibial baseplate component.
Time Frame: 5 years
Population: Knees enrolled in the study.
Measure: Number; unit: Knees
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 180
Number analyzed (Knees) | 181
Knees
  Aseptic Loosening | 5
  Septic Loosening | 9

8. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) Change From Pre-op to Post-op Visits
Description: KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: pre-op, 1, 2, 5 years
Population: Knees with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 179
Number analyzed (Knees) | 180
units on a scale
  KOOS Pain Preoperative: number analyzed (Participants) | 177
  KOOS Pain Preoperative: number analyzed (Knees) | 178
  KOOS Pain Preoperative | 41.51 (18.91)
  KOOS Pain 1 year: number analyzed (Participants) | 146
  KOOS Pain 1 year: number analyzed (Knees) | 147
  KOOS Pain 1 year | 75.09 (21.55)
  KOOS Pain 2 year: number analyzed (Participants) | 134
  KOOS Pain 2 year: number analyzed (Knees) | 134
  KOOS Pain 2 year | 74.67 (21.36)
  KOOS Pain 5 year: number analyzed (Participants) | 93
  KOOS Pain 5 year: number analyzed (Knees) | 93
  KOOS Pain 5 year | 73.95 (21.31)
  KOOS Symptoms Preoperative | 43.39 (18.93)
  KOOS Symptoms 1 year: number analyzed (Participants) | 145
  KOOS Symptoms 1 year: number analyzed (Knees) | 146
  KOOS Symptoms 1 year | 73.02 (21.02)
  KOOS Symptoms 2 year: number analyzed (Participants) | 134
  KOOS Symptoms 2 year: number analyzed (Knees) | 134
  KOOS Symptoms 2 year | 72.95 (19.11)
  KOOS Symptoms 5 year: number analyzed (Participants) | 95
  KOOS Symptoms 5 year: number analyzed (Knees) | 95
  KOOS Symptoms 5 year | 75.88 (17.25)
  KOOS Daily Living Preoperative: number analyzed (Participants) | 177
  KOOS Daily Living Preoperative: number analyzed (Knees) | 178
  KOOS Daily Living Preoperative | 45.56 (20.41)
  KOOS Daily Living 1 year: number analyzed (Participants) | 145
  KOOS Daily Living 1 year: number analyzed (Knees) | 146
  KOOS Daily Living 1 year | 76.43 (21.19)
  KOOS Daily Living 2 year: number analyzed (Participants) | 133
  KOOS Daily Living 2 year: number analyzed (Knees) | 133
  KOOS Daily Living 2 year | 76.17 (21.83)
  KOOS Daily Living 5 year: number analyzed (Participants) | 92
  KOOS Daily Living 5 year: number analyzed (Knees) | 92
  KOOS Daily Living 5 year | 74.99 (20.34)
  KOOS Function Sports and Recreational Preoperative: number analyzed (Participants) | 173
  KOOS Function Sports and Recreational Preoperative: number analyzed (Knees) | 174
  KOOS Function Sports and Recreational Preoperative | 12.56 (19.95)
  KOOS Function Sports and Recreational 1 year: number analyzed (Participants) | 139
  KOOS Function Sports and Recreational 1 year: number analyzed (Knees) | 140
  KOOS Function Sports and Recreational 1 year | 44.10 (34.39)
  KOOS Function Sports and Recreational 2 year: number analyzed (Participants) | 130
  KOOS Function Sports and Recreational 2 year: number analyzed (Knees) | 130
  KOOS Function Sports and Recreational 2 year | 41.86 (33.26)
  KOOS Function Sports and Recreational 5 year: number analyzed (Participants) | 94
  KOOS Function Sports and Recreational 5 year: number analyzed (Knees) | 94
  KOOS Function Sports and Recreational 5 year | 42.77 (43.41)
  KOOS Quality of Life Preoperative | 18.06 (17.90)
  KOOS Quality of Life 1 year: number analyzed (Participants) | 146
  KOOS Quality of Life 1 year: number analyzed (Knees) | 147
  KOOS Quality of Life 1 year | 55.99 (28.20)
  KOOS Quality of Life 2 year: number analyzed (Participants) | 134
  KOOS Quality of Life 2 year: number analyzed (Knees) | 134
  KOOS Quality of Life 2 year | 55.74 (27.71)
  KOOS Quality of Life 5 year: number analyzed (Participants) | 95
  KOOS Quality of Life 5 year: number analyzed (Knees) | 95
  KOOS Quality of Life 5 year | 57.37 (27.56)

9. Secondary Outcome: Hospital Special Surgery (HSS) Patella Score Change From Pre-op to Post-op Visits
Description: The HSS Patella Score incorporates both subjective symptoms and objective data specific to the patellofemoral joint. It consists of one score from 0-100 with a score of 100 indicating no pain, no functional limitations, no tenderness or crepitus and normal quadriceps strength.
Time Frame: pre-op, 1, 2, 5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 170
Number analyzed (Knees) | 171
units on a scale
  HSS Patella Score Preoperative | 45.09 (18.43)
  HSS Patella Score 1 year: number analyzed (Participants) | 142
  HSS Patella Score 1 year: number analyzed (Knees) | 143
  HSS Patella Score 1 year | 76.68 (21.48)
  HSS Patella Score 2 year: number analyzed (Participants) | 128
  HSS Patella Score 2 year: number analyzed (Knees) | 128
  HSS Patella Score 2 year | 80.08 (19.31)
  HSS Patella Score 5 year: number analyzed (Participants) | 87
  HSS Patella Score 5 year: number analyzed (Knees) | 87
  HSS Patella Score 5 year | 78.56 (20.24)

10. Secondary Outcome: Lower Extremity Activity Scale (LEAS) Score Change From Pre-op to Post-op Visits
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: pre-op, 1, 2, 5 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 179
Number analyzed (Knees) | 180
units on a scale
  LEAS Score Preoperative | 7.80 (2.86)
  LEAS Score 1 year: number analyzed (Participants) | 146
  LEAS Score 1 year: number analyzed (Knees) | 147
  LEAS Score 1 year | 9.65 (3.18)
  LEAS Score 2 year: number analyzed (Participants) | 134
  LEAS Score 2 year: number analyzed (Knees) | 134
  LEAS Score 2 year | 9.60 (3.26)
  LEAS Score 5 year: number analyzed (Participants) | 95
  LEAS Score 5 year: number analyzed (Knees) | 95
  LEAS Score 5 year | 9.75 (3.39)

11. Secondary Outcome: Knee Society Score (KSS) Change From Pre-op to Post-op Visits
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, ROM and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: pre-op, 1,2, 5 year
Population: Data based on knees with available data at 1,2 and 5 years postoperative.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Knees
Arm/Group | Triathlon TS Knee
Number analyzed (Participants) | 177
Number analyzed (Knees) | 178
units on a scale
  Pain Motion Mean Preoperative: number analyzed (Participants) | 169
  Pain Motion Mean Preoperative: number analyzed (Knees) | 170
  Pain Motion Mean Preoperative | 39.81 (21.12)
  Pain Motion Mean 1 year: number analyzed (Participants) | 142
  Pain Motion Mean 1 year: number analyzed (Knees) | 143
  Pain Motion Mean 1 year | 85.45 (15.14)
  Pain Motion Mean 2 year: number analyzed (Participants) | 130
  Pain Motion Mean 2 year: number analyzed (Knees) | 130
  Pain Motion Mean 2 year | 83.97 (15.95)
  Pain Motion Mean 5 year: number analyzed (Participants) | 85
  Pain Motion Mean 5 year: number analyzed (Knees) | 85
  Pain Motion Mean 5 year | 82.06 (17.24)
  Function Mean Preoperative | 41.43 (23.09)
  Function Mean 1 year: number analyzed (Participants) | 145
  Function Mean 1 year: number analyzed (Knees) | 146
  Function Mean 1 year | 74.18 (24.00)
  Function Mean 2 year: number analyzed (Participants) | 131
  Function Mean 2 year: number analyzed (Knees) | 131
  Function Mean 2 year | 72.90 (25.12)
  Function Mean 5 year: number analyzed (Participants) | 92
  Function Mean 5 year: number analyzed (Knees) | 92
  Function Mean 5 year | 70.71 (26.51)

ADVERSE EVENTS:
Time Frame: This study requires that all operative site adverse events, regardless of seriousness, and serious systemic adverse events be reported from enrollment through the 5 year postoperative interval. Censored protocol deviations were not included as at risk participants.
Description: Specific Adverse Event terms not used for all Adverse Events.
Groups:
- Operative Adverse Events: Triathlon TS Knee System: Total knee replacement for revision cases
  Operative site events are reported by knee because in the case of bilateral participants (this is when one participant has both knees enrolled in the study), an event can occur in one knee, both knees or the same knee at different times and are counted separately for this reason.
- Non-Operative Adverse Events: Triathlon TS Knee System: Total knee replacement for revision cases
  Non-Operative Site Events are reported by participant.
Arm/Group | Operative Adverse Events | Non-Operative Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/181 | 7/180
Serious Adverse Events (participants affected / at risk) | 37/181 | 40/180
Other Adverse Events (participants affected / at risk) | 59/181 | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=181) | Non-Operative Adverse Events (N=180)
Non-operative Site (Cardiac disorders) | 0/0 (0) | 11 (11)
Non-operative Site (Gastrointestinal disorders) | 0/0 (0) | 5 (5)
Non-operative site (General disorders) | 0/0 (0) | 2 (2)
Operative Site (Infections and infestations) | 15 (17) | 0/0 (0)
Operative Site (Injury, poisoning and procedural complications) | 4 (4) | 0/0 (0)
Non-operative Site (Metabolism and nutrition disorders) | 0/0 (0) | 1 (1)
Non-operative Site (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 10 (14)
Non-operative Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 3 (3)
Non-operative Site (Nervous system disorders) | 0/0 (0) | 2 (2)
Non-operative Site (Psychiatric disorders) | 0/0 (0) | 2 (2)
Non-operative Site (Renal and urinary disorders) | 0/0 (0) | 5 (6)
Non-operative Site (Reproductive system and breast disorders) | 0/0 (0) | 1 (2)
Non-operative Site (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 5 (9)
Non-operative Site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 1 (1)
Non-operative Site (Social circumstances) | 0/0 (0) | 2 (2)
Non-operative Site (Vascular disorders) | 0/0 (0) | 5 (5)
Non-operative Site (Infections and infestations) | 0/0 (0) | 7 (8)
Operative Site (Musculoskeletal and connective tissue disorders) | 24 (25) | 0/0 (0)
Operative Site (Skin and subcutaneous tissue disorders) | 0/0 (0) | 0/0 (0)
Operative Site (Nervous system disorders) | 0/0 (0) | 0/0 (0)
Operative Site (Renal and urinary disorders) | 0/0 (0) | 0/0 (0)
Non-operative Site (Blood and lymphatic system disorders) | 0/0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative Adverse Events (N=181) | Non-Operative Adverse Events (N=180)
Operative Site (Musculoskeletal and connective tissue disorders) | 59 (66) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study.These manuscripts & abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to the submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-03-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT00958789/Prot_SAP_000.pdf
  • Informed Consent Form (2008-04-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT00958789/ICF_001.pdf